CLINICAL TRIAL: NCT03092999
Title: Investigation of Pharmacokinetics, Safety, and Tolerability of Vilaprisan (BAY1002670) in Subjects With Hepatic Impairment (Classified as Child-Pugh A or B) Compared to Sex, Age, and Weight-matched Healthy Subjects Following a Single Oral Dose
Brief Title: Effect of Hepatic Impairment on the Pharmacokinetics, Safety and Tolerability of BAY1002670 (Vilaprisan)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 15251; 2015-005232-18 (EudraCT Number)
Record Dates: First submitted 2017-03-22; First posted 2017-03-28 (Actual); Last update posted 2017-08-18 (Actual); Status verified 2017-07

CONDITIONS: Leiomyoma
Keywords: Pharmacokinetics
MeSH Terms: conditions — Leiomyoma | interventions — vilaprisan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Healthy subjects (Experimental): healthy subjects
  Interventions: Drug: Vilaprisan (BAY1002670)
- Subjects with mild hepatic impairment (Experimental): hepatically impaired patients (classified as Child Pugh A)
  Interventions: Drug: Vilaprisan (BAY1002670)
- Subjects with moderate hepatic impairment (Experimental): hepatically impaired patients (classified as Child Pugh B)
  Interventions: Drug: Vilaprisan (BAY1002670)

INTERVENTIONS:
Drug: Vilaprisan (BAY1002670) — 2 mg tablet, single dose, oral administration

SUMMARY:
Evaluate the potential effect of hepatic impairment on the pharmacokinetics, safety and tolerability of BAY1002670 (vilaprisan)

ELIGIBILITY:
Inclusion Criteria:

For all subjects:

* The informed consent must be signed before any study specific tests or procedures are done
* White/Caucasian men and women aged between 18 to 79 years (inclusive )
* Body mass index (BMI): 18 to 34 kg/m2 (both inclusive)
* Ability to understand and follow study-related instructions
* Women and men of reproductive potential must agree to use adequate contraception when sexually active. This applies for the time period between signing of the informed consent form and three months after administration of study drug. Subjects must agree to use two non-hormonal methods for contraception simultaneously (e.g. condom or diaphragm, plus spermicide) throughout the study when sexually active.

This is not required if safe contraception is achieved by a permanent method, such as hysterectomy, bilateral fallopian tube ligation or vasectomy.

For subjects with hepatic impairment:

* Subjects with documented liver cirrhosis confirmed by histopathology, laparoscopy, fibroscan, or ultrasound
* Subjects with hepatic impairment (Child-Pugh A or B)
* Subjects with stable liver disease, i.e. same Child-Pugh class in the last 2 months

Exclusion Criteria:

* Any relevant disease within 4 weeks prior to study drug administration requiring medical treatment
* Known severe allergies, non-allergic drug reactions, or multiple drug allergies
* Use containing sex hormones within 4 weeks to six months before first study drug administration
* Use of CYP3A4 and P-glycoprotein inhibitors or inducers
* Use of drugs which may affect absorption
* Major change of medication <2 weeks prior study drug administration
* Deviations from normal range in physical examination, gynecological examination, clinical chemistry, hematology, or urinalysis considered to be relevant by the investigator
* Any criteria which, in the opinion of the investigator, make study participation unadvisable for scientific, compliance, safety, or medical reasons

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2017-03-28 (Actual); Primary Completion 2017-07-17 (Actual); Study Completion 2017-07-17 (Actual)

PRIMARY OUTCOMES:
Area under the concentration vs. time curve in plasma from zero to infinity (AUCu) (unbound) | At pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16 hours and at 1, 2, 3, 7, 10, 13, 16, 20 days
  Exposure of Vilaprisan in plasma following a single dose administration
Maximum observed (unbound) drug concentration (Cmax,u) | At pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16 hours and at 1, 2, 3, 7, 10, 13, 16, 20 days
  Maximum observed (unbound) drug concentration (Cmax,u) in measured matrix after a single dose administration

SECONDARY OUTCOMES:
Frequency of Treatment Emergent Adverse Events | Up to 20 days
  Frequency of Treatment Emergent Adverse Events as a measure of safety and tolerability
Severity of Treatment Emergent Adverse Events | Up to 20 days
  The intensity of an AE is classified according to the following categories:
  * Mild
  * Moderate
  * Severe
Changes in blood laboratory parameters | Up to 20 days
  Changes in blood laboratory parameters including hematology, clotting status, serum chemistry
Changes in urine laboratory parameters | Up to 20 days
  Changes in urine laboratory parameters including urine analysis, urine pregnancy tests
Changes in Vital Signs | Up to 20 days
  Changes in Vital Signs, including blood pressure, pulse, body temperature
Changes in Electrocardiogram (ECG) | Up to 20 days
  ECG (12-lead) after ≥10 minutes supine rest

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (2):
- Germany (2):
  - CRS Clinical-Research-Services Kiel GmbH, Kiel, Schleswig-Holstein
  - Universitätsklinikum Schleswig-Holstein / AÖR, Lübeck